CLINICAL TRIAL: NCT00326781
Title: Bio-Behavioral Predictors of the Efficacy of Nicotine Replacement Therapy - Transdisciplinary Tobacco Use Research Center (TTURC), Project 2
Brief Title: Bio-Behavioral Predictors of the Efficacy of Nicotine Replacement Therapy (NRT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Caryn Lerman, Ph.D., University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 703294; P50CA084718 (NIH)
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2010-03-19 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-03

CONDITIONS: Smoking
Keywords: Nicotine nasal spray + counseling; Transdermal nicotine + counseling
MeSH Terms: conditions — Smoking | interventions — Nicotine; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Nasal Spray (Active Comparator)
  Interventions: Drug: Nicotine Nasal Spray
- Transdermal Nicotine patch (Active Comparator)
  Interventions: Drug: Nicoderm Transdermal Patch

INTERVENTIONS:
Drug: Nicoderm Transdermal Patch — The dosing schedule is as follows: 4 weeks of 21mg per 24 hours, 2 weeks of 14mg per 24 hours, and 2 weeks of 7mg per 24 hours. Treatment lasted 8 weeks.
  Other Names: Nicoderm®
  Arms: Transdermal Nicotine patch
Drug: Nicotine Nasal Spray — 8 weeks of self-administered nicotine nasal spray at 40 recommended doses per day, tapering by 1/3 for the last 4 weeks. Nasal spray dosing was 0.5 mg spray per nostril (1 mg) for a maximum of 5 doses per hour and 40 doses per day. This dosing schedule is based on the average nicotine intake per cigarette of 1 mg per cigarette. Treatment lasted 8 weeks.
  Other Names: Nicotrol
  Arms: Nicotine Nasal Spray

SUMMARY:
The purpose of this research study is to:

1. compare the effectiveness of a nicotine patch and nicotine nasal spray for smoking cessation; and
2. identify predictors of response to these alternate forms of nicotine replacement therapy (NRT).

DETAILED DESCRIPTION:
The ultimate objective is to obtain information necessary to match NRT to those smokers with the greatest need and likelihood of benefit. The investigators hypothesize that the nicotine nasal spray (NS) will result in significantly higher abstinence rates than transdermal nicotine (TN) for the following subgroups of smokers: those with genotypes associated with less transmission of dopamine or serotonin, or greater metabolism of nicotine; and those with higher levels of novelty-seeking, depression, and attention deficit symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be male and female smokers age 18-75.
* Eligible smokers will be those currently smoking at least 10 cigarettes a day.

Exclusion Criteria:

* Planning a pregnancy, pregnant, or lactating
* Current addiction to opiates, cocaine, or stimulants
* Skin allergies or chronic dermatitis (based on medical history/self-report)
* An Axis 1 major psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 1999-12; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Munafo MR, Johnstone EC, Wileyto EP, Shields PG, Elliot KM, Lerman C. Lack of association of 5-HTTLPR genotype with smoking cessation in a nicotine replacement therapy randomized trial. Cancer Epidemiol Biomarkers Prev. 2006 Feb;15(2):398-400. doi: 10.1158/1055-9965.EPI-05-0648. No abstract available. PMID 16492936
- [Result] Malaiyandi V, Lerman C, Benowitz NL, Jepson C, Patterson F, Tyndale RF. Impact of CYP2A6 genotype on pretreatment smoking behaviour and nicotine levels from and usage of nicotine replacement therapy. Mol Psychiatry. 2006 Apr;11(4):400-9. doi: 10.1038/sj.mp.4001794. PMID 16402128
- [Result] Dahl JP, Jepson C, Levenson R, Wileyto EP, Patterson F, Berrettini WH, Lerman C. Interaction between variation in the D2 dopamine receptor (DRD2) and the neuronal calcium sensor-1 (FREQ) genes in predicting response to nicotine replacement therapy for tobacco dependence. Pharmacogenomics J. 2006 May-Jun;6(3):194-9. doi: 10.1038/sj.tpj.6500358. PMID 16402081
- [Result] Lerman C, Jepson C, Wileyto EP, Epstein LH, Rukstalis M, Patterson F, Kaufmann V, Restine S, Hawk L, Niaura R, Berrettini W. Role of functional genetic variation in the dopamine D2 receptor (DRD2) in response to bupropion and nicotine replacement therapy for tobacco dependence: results of two randomized clinical trials. Neuropsychopharmacology. 2006 Jan;31(1):231-42. doi: 10.1038/sj.npp.1300861. PMID 16123753
- [Result] Rukstalis M, Jepson C, Patterson F, Lerman C. Increases in hyperactive-impulsive symptoms predict relapse among smokers in nicotine replacement therapy. J Subst Abuse Treat. 2005 Jun;28(4):297-304. doi: 10.1016/j.jsat.2005.02.002. PMID 15925263
- [Result] Colilla S, Lerman C, Shields PG, Jepson C, Rukstalis M, Berlin J, DeMichele A, Bunin G, Strom BL, Rebbeck TR. Association of catechol-O-methyltransferase with smoking cessation in two independent studies of women. Pharmacogenet Genomics. 2005 Jun;15(6):393-8. doi: 10.1097/01213011-200506000-00004. PMID 15900212
- [Result] Strasser AA, Kaufmann V, Jepson C, Perkins KA, Pickworth WB, Wileyto EP, Rukstalis M, Audrain-McGovern J, Lerman C. Effects of different nicotine replacement therapies on postcessation psychological responses. Addict Behav. 2005 Jan;30(1):9-17. doi: 10.1016/j.addbeh.2004.04.005. PMID 15561445
- [Result] Strasser AA, Pickworth WB, Patterson F, Lerman C. Smoking topography predicts abstinence following treatment with nicotine replacement therapy. Cancer Epidemiol Biomarkers Prev. 2004 Nov;13(11 Pt 1):1800-4. PMID 15533910
- [Result] Lerman C, Kaufmann V, Rukstalis M, Patterson F, Perkins K, Audrain-McGovern J, Benowitz N. Individualizing nicotine replacement therapy for the treatment of tobacco dependence: a randomized trial. Ann Intern Med. 2004 Mar 16;140(6):426-33. doi: 10.7326/0003-4819-140-6-200403160-00009. PMID 15023708
- [Result] Lerman C, Wileyto EP, Patterson F, Rukstalis M, Audrain-McGovern J, Restine S, Shields PG, Kaufmann V, Redden D, Benowitz N, Berrettini WH. The functional mu opioid receptor (OPRM1) Asn40Asp variant predicts short-term response to nicotine replacement therapy in a clinical trial. Pharmacogenomics J. 2004;4(3):184-92. doi: 10.1038/sj.tpj.6500238. PMID 15007373
- [Result] Patterson F, Jepson C, Kaufmann V, Rukstalis M, Audrain-McGovern J, Kucharski S, Lerman C. Predictors of attendance in a randomized clinical trial of nicotine replacement therapy with behavioral counseling. Drug Alcohol Depend. 2003 Nov 24;72(2):123-31. doi: 10.1016/s0376-8716(03)00194-7. PMID 14636967
- [Result] Lerman C, Caporaso N, Main D, Audrain J, Boyd NR, Bowman ED, Shields PG. Depression and self-medication with nicotine: the modifying influence of the dopamine D4 receptor gene. Health Psychol. 1998 Jan;17(1):56-62. doi: 10.1037//0278-6133.17.1.56. PMID 9459071
- [Derived] Ashare RL, Wileyto EP, Perkins KA, Schnoll RA. The first 7 days of a quit attempt predicts relapse: validation of a measure for screening medications for nicotine dependence. J Addict Med. 2013 Jul-Aug;7(4):249-54. doi: 10.1097/ADM.0b013e31829363e1. PMID 23669629
- [Derived] Javitz HS, Lerman C, Swan GE. Comparative dynamics of four smoking withdrawal symptom scales. Addiction. 2012 Aug;107(8):1501-11. doi: 10.1111/j.1360-0443.2012.03838.x. Epub 2012 Apr 17. PMID 22321019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between December 1999 and July 2003.
Groups:
- Transdermal Nicotine: Half of randomized participants received 8-weeks of transdermal nicotine (Nicoderm CQ). The dosing schedule was as follows: 4 weeks of 21mg per 24 hours, 2 weeks of 14mg per 24 hours, and 2 weeks of 7mg per 24 hours.
- Nicotine Nasal Spray: Half of all participants received nicotine nasal spray. 8 weeks of self-administered nicotine nasal spray @ 40 recommended doses per day, tapering by 1/3 for the last 4 weeks. Nasal spray dosing was 0.5 mg spray per nostril (1 mg) for a maximum of 5 doses per hour and 40 doses per day. This dosing schedule is based on the average nicotine intake per cigarette of 1 mg per cigarette.
Period: Overall Study
Arm/Group | Transdermal Nicotine | Nicotine Nasal Spray
Started | 344 | 330
Completed | 302 | 298
Not Completed | 42 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Nicotine | Nicotine Nasal Spray | Total
Number analyzed (Participants) | 344 | 330 | 674
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 329 | 321 | 650
  >=65 years | 15 | 9 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 45.63 (10.88) | 45.41 (10.37) | 45.53 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 185 | 359
  Male | 170 | 145 | 315
Region of Enrollment [Number; unit: participants]
  United States | 344 | 330 | 674

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence at End of Treatment (Self-report)(Defined as the Number of Consecutive Days Without Smoking a Cigarette for Each Subject)
Description: A self-report measure of continuous abstinence at end of treatment. It is defined as the number of consecutive days without smoking a cigarette for each subject, as determined by the Timeline Followback (TLFB), completed by research staff. The TLFB is an assessment tool that obtains estimates of daily smoking. Using a calendar, people provide retrospective estimates of their daily smoking over a specified time period that can vary up to 12 months from the interview date. The TLFB has also been used to assess other forms of substance abuse (e.g., alcohol, drugs, etc.).
Time Frame: End of Treatment (8-weeks after quit date)
Population: Analysis was intention to treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Transdermal Nicotine | Nicotine Nasal Spray
Number analyzed (Participants) | 344 | 330
Participants | 83 | 75

2. Secondary Outcome: Verified 7-day Point Prevalence Abstinence at End Of Treatment.
Description: End-of-Treatment (EOT) is defined as the phone survey that takes place at the end of each subject's nicotine replacement therapy treatment. The EOT took place up to 8 weeks after participants began the study and also utilized the Timeline Followback. It is a 7-day point prevalence measure describing a subject's ability to remain abstinent from smoking for the 7 previous days occurring before a subject's EOT phone survey.
  This was verified by a Carbon Monoxide breath reading taking place within a week of a subject's End of Treatment phone survey.
Time Frame: End of Treatment
Measure: Number; unit: participants
Arm/Group | Transdermal Nicotine | Nicotine Nasal Spray
Number analyzed (Participants) | 344 | 330
participants | 112 | 95

ADVERSE EVENTS:
Arm/Group | Transdermal Nicotine | Nicotine Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/344 | 0/330
Other Adverse Events (participants affected / at risk) | 0/344 | 0/330

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No